CLINICAL TRIAL: NCT02970071
Title: The Application Value of STIC in the Diagnosis of Fetal Complex Congenital Heart Disease
Acronym: STIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-16-036
Record Dates: First submitted 2016-11-18; First posted 2016-11-21 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-09

CONDITIONS: Congenital Heart Disease
Keywords: Spatio-Temporal Image Correlation; Complicated congenital heart disease; Echocardiography
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Fetal congenital heart disease cases: Gravidas with fetal congenital heart disease diagnosed by fetal echocardiography

SUMMARY:
The objective of this study is to use of STIC technology to assist the traditional echocardiography to diagnose the fetal congenital heart disease accurately and then to provide a basis for prenatal counseling.

DETAILED DESCRIPTION:
This is a diagnostic test in Shanghai Xinhua hospital from Nov.2016 to Dec.2017. 265 Cases are gravidas with fetal congenital heart disease diagnosed by echocardiography.Only gravidas who are willing to have complete pregnancy checks and finally delivery or abortion in the hospital are interviewed are eligible for the study. Study participants will be asked for their informed consent.We collect their fetal 2D echocardiography and STIC images every 4-6 weeks during pregnancy and 1 weeks after the baby giving birth we finish their neonatal echocardiography.

ELIGIBILITY:
Inclusion Criteria:

1. Gravida with singleton pregnancy taking fetal echocardiography.
2. No virus infection or drug use history, no harmful substances in the early pregnancy.
3. Complete pregnancy check in the hospital, and finally delivery or abortion in the hospital.
4. On the basis of informed consent，willing to cooperate with our group.

Exclusion Criteria:

1. Elderly pregnant women (>35 years old)
2. Twin or multiple pregnancy
3. Pregnant women suffering from mental illness, can't take care of themselves.
4. Fetus diagnosed with other abnormalities (except congenital heart defects)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Gravidas with singleton pregnancy living in SHANGHAI
Sampling Method: Non-Probability Sample
Enrollment: 265 (Estimated)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Fetal Congenital heart disease | Nov 2016 to Dec 2018
  If an enrolled gravida chooses to terminate her pregnancy, autopsy confirmation will be performed ;If the gravida continues her pregnancy, the outcome will be measured by neonatal echocardiography or surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Xinhua Hospital Shanghai Jiao Tong University School of Medicine, Principal Investigator — Investigator
Locations (1):
- Xinhua Hospital,Shanghai Jiao Tong University School of Medicine, Yangpu, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wren C, Reinhardt Z, Khawaja K. Twenty-year trends in diagnosis of life-threatening neonatal cardiovascular malformations. Arch Dis Child Fetal Neonatal Ed. 2008 Jan;93(1):F33-5. doi: 10.1136/adc.2007.119032. Epub 2007 Jun 7. PMID 17556383
- [Result] Kim N, Friedberg MK, Silverman NH. Diagnosis and prognosis of fetuses with double outlet right ventricle. Prenat Diagn. 2006 Aug;26(8):740-5. doi: 10.1002/pd.1500. PMID 16807954
- [Result] DeVore GR, Falkensammer P, Sklansky MS, Platt LD. Spatio-temporal image correlation (STIC): new technology for evaluation of the fetal heart. Ultrasound Obstet Gynecol. 2003 Oct;22(4):380-7. doi: 10.1002/uog.217. PMID 14528474